CLINICAL TRIAL: NCT04206813
Title: An Open-Label Clinical Trial Evaluating the Immunogenicity of the 9vHPV Vaccination Regimen Over 6 Months Among Women Aged 16 to 45 Years Old, An Exploratory Immunogenicity Study
Brief Title: An Exploratory Open-Label Clinical Trial Evaluating the Immunogenicity of the 9-valent 2-dose HPV Vaccination Regimen
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H-39051
Record Dates: First submitted 2019-12-15; First posted 2019-12-20 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: HPV Infection
Keywords: Gardasil; Immunogenicity; 9-valent 2-dose HPV vaccination; 9-valent 3-dose HPV vaccination
MeSH Terms: conditions — Papillomavirus Infections | interventions — Human Papillomavirus Recombinant Vaccine nonavalent; Clinical Protocols

STUDY DESIGN:
Intervention Model Description: The control group will have 120 subjects will receive a 3-dose regimen as recommended by Center for Disease Control (CDC) given at 0, 2 and 6 months. The intervention group will have 240 subjects who will receive a modified 3-dose regimen given at 0, 6, and 12 months. Both groups will have HPV titers drawn at Visit 1 (pre-vaccination) and Visit 7 (after three doses for the Control group and 2 doses for the Intervention group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention group (Experimental): 240 eligible women will receive a 2-dose regimen of Gardasil 9 at (0 and 6 months, followed by a rescue 3rd dose at month 12)
  Interventions: Drug: Gardasil 9 2 dose regimen; Drug: Gardasil 9 rescue dose
- Control group (Active Comparator): 120 eligible women will receive the standard 3-dose regimen of Gardasil 9 at (0, 2, 6 months)
  Interventions: Drug: Gardasil 9 3 dose regimen

INTERVENTIONS:
Drug: Gardasil 9 2 dose regimen — a 2-dose regimen of Gardasil 9 at 0 and 6 months
  Other Names: Human Papillomavirus 9-valent Vaccine, Recombinant
  Arms: Intervention group
Drug: Gardasil 9 3 dose regimen — standard 3-dose regimen of Gardasil 9 at 0, 2, 6 months
  Other Names: Human Papillomavirus 9-valent Vaccine, Recombinant
  Arms: Control group
Drug: Gardasil 9 rescue dose — A rescue dose of Gardasil 9 will be given at 12 months
  Other Names: Human Papillomavirus 9-valent Vaccine, Recombinant
  Arms: Intervention group

SUMMARY:
The goal of this study is to explore and evaluate whether a 2-dose schedule of Gardasil 9 among young and mid-adult women 16-45 years of age is generally safe and immunogenic, with an antibody response that is not inferior to that observed of a 3-dose schedule of Gardasil 9 among women aged 16-26 years old. The investigators thought that having a 2-dose vaccination regimen for individuals 16 to 45 would provide a more robust dataset than those of 27 to 45 years old.

DETAILED DESCRIPTION:
The investigators will identify potential eligible subjects from the Boston Medical Center (BMC) Clinical Data Warehouse from the following BMC clinics: Pediatrics, Adolescent Medicine, Family Medicine, Obstetric/ Gynecology (OB/GYN), and Women's Health/Adult Primary Care. The research team will mail a recruitment opt-out letter signed by the principal investigator to the participant along with a study flyer. The recruitment letter will inform the participant that a research member may contact them via phone within two week to provide more information regarding the study.

Participants opting-in will be called and interviewed with the study recruitment script and eligibility will be determined. Eligible participants who agree to participate (in-person or over the phone), will be scheduled to come to the Boston University (BU) General Clinical Research Unit (GCRU) to complete the consent process. At the baseline visit participants will be assigned into the appropriate group (control vs. intervention) based on their age.

ELIGIBILITY:
Inclusion Criteria:

* Women receiving care at Boston Medical Center

Exclusion Criteria:

* Currently pregnant
* Prior HPV vaccination
* A history of severe allergic reaction, including known allergy to any vaccine component, specially severe allergic to yeast
* Immunocompromised/previous immunosuppressive therapy
* Thrombocytopenia or other coagulation disorder
* Currently breastfeeding

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 352 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in immunogenicity of Gardasil 9 | baseline and 7 months
  Immunogenicity will be measured by serum antibodies assessed by ELISA to the nine HPV types (anti-HPV 6/11/16/18/31/33/45/ 52/58 where positive anti-HPV serum levels are defined as >30, >16, >20, >24, >10, >8, >8, >8, or >8 milli Merck units (mMU)/mL respectively).
Change in geometric mean titers ratios | baseline and 7 months
  The geometric mean titers (GMT) ratios will be determined by a post-vaccination geometric mean titer (GMT) ratio with a pre-stated analysis of variance model (95% Confidence Interval lower bound >0.5).

SECONDARY OUTCOMES:
Number of participants with HPV seropositivity at day 1 | day 1
  The number of participant who test positive in mili Unit (nMU) which will be will be defined as anti-HPV 6/11/16/18/31/33/45/ 52/58 positive if her anti-HPV serum level is >30, >16, >20, >24, >10, >8, >8, >8, or >8 milli Merck units (mMU)/mL for the 9 types, respectively. The serum testing will be under the direction of Merck research lab.
Number of participants with HPV seropositivity at month 7 | month 7
  The number of participant who test positive in mili Unit (nMU) which will be will be defined as anti-HPV 6/11/16/18/31/33/45/ 52/58 positive if her anti-HPV serum level is >30, >16, >20, >24, >10, >8, >8, >8, or >8 milli Merck units (mMU)/mL for the 9 types, respectively. The serum testing will be under the direction of Merck research lab.

CONTACTS AND LOCATIONS:
Overall Officials: Carl G Streed, MD MPH, Principal Investigator — Boston Medical Center, Internal Medicine
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meites E, Kempe A, Markowitz LE. Use of a 2-Dose Schedule for Human Papillomavirus Vaccination - Updated Recommendations of the Advisory Committee on Immunization Practices. MMWR Morb Mortal Wkly Rep. 2016 Dec 16;65(49):1405-1408. doi: 10.15585/mmwr.mm6549a5. PMID 27977643
- [Background] Joura EA, Giuliano AR, Iversen OE, Bouchard C, Mao C, Mehlsen J, Moreira ED Jr, Ngan Y, Petersen LK, Lazcano-Ponce E, Pitisuttithum P, Restrepo JA, Stuart G, Woelber L, Yang YC, Cuzick J, Garland SM, Huh W, Kjaer SK, Bautista OM, Chan IS, Chen J, Gesser R, Moeller E, Ritter M, Vuocolo S, Luxembourg A; Broad Spectrum HPV Vaccine Study. A 9-valent HPV vaccine against infection and intraepithelial neoplasia in women. N Engl J Med. 2015 Feb 19;372(8):711-23. doi: 10.1056/NEJMoa1405044. PMID 25693011
- [Background] Castellsague X, Munoz N, Pitisuttithum P, Ferris D, Monsonego J, Ault K, Luna J, Myers E, Mallary S, Bautista OM, Bryan J, Vuocolo S, Haupt RM, Saah A. End-of-study safety, immunogenicity, and efficacy of quadrivalent HPV (types 6, 11, 16, 18) recombinant vaccine in adult women 24-45 years of age. Br J Cancer. 2011 Jun 28;105(1):28-37. doi: 10.1038/bjc.2011.185. Epub 2011 May 31. PMID 21629249
- [Background] Giuliano AR, Isaacs-Soriano K, Torres BN, Abrahamsen M, Ingles DJ, Sirak BA, Quiterio M, Lazcano-Ponce E. Immunogenicity and safety of Gardasil among mid-adult aged men (27-45 years)--The MAM Study. Vaccine. 2015 Oct 13;33(42):5640-5646. doi: 10.1016/j.vaccine.2015.08.072. Epub 2015 Sep 4. PMID 26343499
- [Background] Romanowski B, Schwarz TF, Ferguson LM, Peters K, Dionne M, Schulze K, Ramjattan B, Hillemanns P, Catteau G, Dobbelaere K, Schuind A, Descamps D. Immunogenicity and safety of the HPV-16/18 AS04-adjuvanted vaccine administered as a 2-dose schedule compared with the licensed 3-dose schedule: results from a randomized study. Hum Vaccin. 2011 Dec;7(12):1374-86. doi: 10.4161/hv.7.12.18322. Epub 2011 Dec 1. PMID 22048171
- [Background] Basu P, Muwonge R, Bhatla N, Nene BM, Joshi S, Esmy PO, Poli URR, Joshi G, Verma Y, Zomawia E, Shastri SS, Pimple S, Anantharaman D, Prabhu PR, Hingmire S, Sauvaget C, Lucas E, Pawlita M, Gheit T, Jayant K, Malvi SG, Siddiqi M, Michel A, Butt J, Sankaran S, Rameshwari Ammal Kannan TP, Varghese R, Divate U, Willhauck-Fleckenstein M, Waterboer T, Muller M, Sehr P, Vashist S, Mishra G, Jadhav R, Thorat R, Tommasino M, Pillai MR, Sankaranarayanan R; Indian HPV vaccine study group. Two-dose recommendation for Human Papillomavirus vaccine can be extended up to 18 years - updated evidence from Indian follow-up cohort study. Papillomavirus Res. 2019 Jun;7:75-81. doi: 10.1016/j.pvr.2019.01.004. Epub 2019 Jan 31. PMID 30711698
- [Background] Meites E, Szilagyi PG, Chesson HW, Unger ER, Romero JR, Markowitz LE. Human Papillomavirus Vaccination for Adults: Updated Recommendations of the Advisory Committee on Immunization Practices. MMWR Morb Mortal Wkly Rep. 2019 Aug 16;68(32):698-702. doi: 10.15585/mmwr.mm6832a3. PMID 31415491
- [Background] Hernandez-Avila M, Torres-Ibarra L, Stanley M, Salmeron J, Cruz-Valdez A, Munoz N, Herrero R, Villasenor-Ruiz IF, Lazcano-Ponce E. Evaluation of the immunogenicity of the quadrivalent HPV vaccine using 2 versus 3 doses at month 21: An epidemiological surveillance mechanism for alternate vaccination schemes. Hum Vaccin Immunother. 2016;12(1):30-8. doi: 10.1080/21645515.2015.1058458. Epub 2015 Jul 25. PMID 26211489
- [Background] Block SL, Nolan T, Sattler C, Barr E, Giacoletti KE, Marchant CD, Castellsague X, Rusche SA, Lukac S, Bryan JT, Cavanaugh PF Jr, Reisinger KS; Protocol 016 Study Group. Comparison of the immunogenicity and reactogenicity of a prophylactic quadrivalent human papillomavirus (types 6, 11, 16, and 18) L1 virus-like particle vaccine in male and female adolescents and young adult women. Pediatrics. 2006 Nov;118(5):2135-45. doi: 10.1542/peds.2006-0461. PMID 17079588
- [Background] Van Damme P, Olsson SE, Block S, Castellsague X, Gray GE, Herrera T, Huang LM, Kim DS, Pitisuttithum P, Chen J, Christiano S, Maansson R, Moeller E, Sun X, Vuocolo S, Luxembourg A. Immunogenicity and Safety of a 9-Valent HPV Vaccine. Pediatrics. 2015 Jul;136(1):e28-39. doi: 10.1542/peds.2014-3745. PMID 26101366
- [Background] Yifan Huang, Jason C. Hsu, Hochberg's Step-Up Method: Cutting Corners Off Holm's Step-Down Method, Biometrika, Volume 94, Issue 4, December 2007, Pages 965-975, https://doi.org/10.1093/biomet/asm067
- See also: Centers for Disease Control and Prevention, Human Papillomavirus (HPV) facts. — https://www.cdc.gov/sti/about/about-genital-hpv-infection.html
- See also: Centers for Disease Control and Prevention, on how many cancers are linked with HPV each year. — https://www.cdc.gov/cancer/hpv/
- See also: Merck Sharp & Dohme Corp. An Open-Label Phase III Clinical Trial to Study the Immunogenicity and Tolerability of GARDASIL®9 (A Multivalent Human Papillomavirus [HPV] L1 Virus-Like Particle Vaccine) in Adult Women Compared to Young Adult Women — http://clinicaltrials.gov/ct2/show/study/NCT03158220
- See also: Food and Drug Administration. Prescribing information [package insert]. Gardasil 9 (human papillomavirus 9-valent vaccine, recombinant). — https://www.fda.gov/media/90064/download
- See also: Luxembourg A. 9vHPV immunogenicity and safety trial in mid-adult females. Advisory Committee on Immunization Practices (ACIP). — https://www.cdc.gov/acip/?CDC_AAref_Val=https://www.cdc.gov/vaccines/acip/meetings/downloads/slides-2019-06/HPV-3-Luxembourg-508.pdf
- See also: Implementing Constrained or Balanced-Across-the-Centers Randomization with SAS v8 Procedure PLAN Song CQ. — https://www.lexjansen.com/pharmasug/2003/StatisticsPharmacokinetics/sp007.pdf